CLINICAL TRIAL: NCT05290025
Title: Integration of Smoking Cessation Into Standard Treatment for People Receiving Opioid Agonist Therapy Who Are Smoking Tobacco: Protocol for a Randomised Controlled Trial
Brief Title: Easy Access to Smoking Cessation for People Receiving Opioid Agonist Therapy Who Are Smoking Tobacco
Acronym: BAReNikotin
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Stavanger HF (Other Government); Helse Vest (Other); University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 155386/ REK-B
Record Dates: First submitted 2022-01-31; First posted 2022-03-22 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Smoking Cessation; Substance-Related Disorders
Keywords: Tobacco Use Cessation Devices; Smoking Cessation; Opioid-Related Disorders; Opiate Substitution Treatment
MeSH Terms: conditions — Smoking Cessation; Substance-Related Disorders; Opioid-Related Disorders | interventions — Tobacco Use Cessation Devices; Nicotine Chewing Gum; Mass Screening

STUDY DESIGN:
Intervention Model Description: Participants randomised to the intervention arm will receive an individually tailored plan for smoking cessation or reduction of number of cigarettes smoked. Smoking cessation treamtent consist of brief behavoiural interventions and provision of prescription-free nicotin patches, nicotine lozenges or nicotine gum.
  Participants will collect the medication for smoking cessation once a week in parallel with delivery of OAT medication. Medication is individually packed for each patient and one week's use. Staff handing out the medication will give the patients a brief intervention asking about how they are progressing in their smoking cessation attempt, how much the patient smoked the day before and if they took the medication as planned. At mid of the intervention period around week 16 (12-20 weeks after intervention initiation), treatment effect measures will be collected
Who Masked: Outcomes Assessor
Masking Description: Even though complete blinding is regarded as difficult and infeasible, patients will be informed of the follow-up they will receive but not on other follow-up alternatives that are used or the exact hypotheses for the study. Outcomes assessor will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients will be offered brief weekly behavioural interventions for smoking cessation and prescription-free nicotine replacement products in addidition standard opioid replacement therapy.
  Interventions: Drug: Nicotine patch; Drug: Nicotine gum; Drug: Nicotine lozenge; Behavioral: Smoking cessation counselling; Other: Screening for use of tobacco products; Other: Screening for interest in smoking cessation
- Intitial screening only (Other): Participants will receive standard opioid replacement therapy. At the start of the intervention number of cigarettes smoked during the past week will be recorded. Smokers will be adviced to make a cessation or reduction attempt. Advice that nicotine replacement products ( patches, lozenges or gum) may be bought over the counter in grocery-stores and pharmacies and information about goverment home-pages giving cessation advice.
  Interventions: Other: Screening for use of tobacco products; Other: Screening for interest in smoking cessation

INTERVENTIONS:
Drug: Nicotine patch — > 20 cigarettes per day: 21 mg nicotine/ 24 hours 10-20 cigarettes per day: 14 mg nicotine/ 24 hours 5-10 cigarettes per day: 7 mg nicotine/ 24 hours
  Arms: Intervention
Drug: Nicotine gum — Nicotine chewing gum will be available in 1 and 2 mg strengths. Patients may individually choose which strength to use. Maximum 12 chewing gums per day
  Arms: Intervention
Drug: Nicotine lozenge — Nicotine lozenges will be available in 1 and 2 mg strengths. Patients may individually choose which strength to use. Maximum 12 lozenges per day
  Arms: Intervention
Behavioral: Smoking cessation counselling — Once a week patients are asked about progress in cessation attempt. Sigaretts smoked the last week are recorded. Goal is set for the next week. Information on typical nicotine withdrawal symptoms and ameliorating techniques.
  Arms: Intervention
Other: Screening for use of tobacco products — At the initiation of the trial screening questions about cigarett use for the last day and week.
Other: Screening for interest in smoking cessation — At the initiation of the trial all smoking participants are asked if the are interested in changing their smoking habits. They are given three alternatives: will make cessation attempt; will make reduction attempt; not certain.

SUMMARY:
Background: About 85% of those receiving opioid agonist therapy (OAT) for opioid dependence are smoking tobacco. Cigarette smoke lead to lunge diseases and cause illness and death within this group. BAReNikotin is a multicentre randomised controlled clinical trial that will test if integration of smoking cessation therapy to clinical practice at OAT-clinics will increase the rate of OAT-patients that quit smoking.

Intervention: The patients selected for the intervention arm will receive smoking cessation therapy including weekly brief behavioural interventions and prescription-free nicotine replacement products such as nicotine lozenges, patches and chewing gum for at least 16 weeks. This will be compared to a group of patients, who does not receive any help to quit smoking, apart from intial screening of smoking behaviour and advice on where to buy nicotine replacement products.

The patients will have to attend OAT outpatient clinics in Bergen and Stavanger, Norway. The main evaluation will take place 16 weeks after the start of the study.

Study population: The target group will be patients with severe opioid dependence receiving OAT from outpatient clinics in the aforementioned cities who are smoking tobacco daily.

Expected outcome: The primary goal of the study is to see how many of those patients that are offered smoking cessation treatment, that have stopped smoking or reduced the number of cigarettes smoked by at least one half by the end of the intervention. We will also investigate if quitting smoking changes the well-being, physical fitness and quality of life of the participants. If the nicotine replacement therapy is safe and efficacious, it can be considered for further scale-up.

DETAILED DESCRIPTION:
Background: About 85% of those receiving opioid agonist therapy (OAT) for opioid dependence are smoking tobacco. Smoke-related pulmonary diseases are significant contributors to morbidity and mortality within this group. BAReNikotin is a multicentre randomised controlled clinical trial that will compare if integrated smoking cessation therapy increases the rate om smoking cessation compared to standard treatment at OAT-clinics among patients who receive OAT.

Study design: BAReNikotin is a multicentre, randomised controlled clinical trial that will recruit 266 patients receiving OAT in Bergen and Stavanger, Norway.

Intervention: The patients selected for the intervention arm will receive smoking cessation therapy including weekly brief behavioural interventions and prescription-free nicotine replacement products such as nicotine lozenges, patches and chewing gum for at least 16 weeks. This will be compared to a group of patients, who does not receive any help to quit smoking, apart from intial screening of smoking behaviour and advice on where to buy nicotine replacement products.

Study population: The target group will be patients with severe opioid dependence receiving OAT from outpatient clinics in the aforementioned cities who are smoking tobacco daily.

Expected outcome: The primary outcomes are smoking cessation verified by carbon monoxide (CO)-levels or at least a 50 % reduction in the number of cigarettes smoked. The study will assess changes in psychological well-being, impact of smoking cessation and reduction on inflammation, changes in physical health relative, quality of life and fatigue. If the integraded approach increases the number of successful cessation attempts this would be a strong argument for including smoking cessation therapy into regulart OAT-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Receiving OAT from an included outpatient clinic with weekly follow-up
* Smoking at least one cigarette per day or seven cigarettes per week
* Obtaining informed consent

Exclusion Criteria:

* Allergies or prior anaphylactic reactions to medication used
* Smoking less than three times a week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Smoking cessation | Mid of the intervention period 16 weeks after initiation
  Smoking cessation verified by CO-levels below 6 at the end of the intervention
Smoking reduction | Mid of the intervention period 16 weeks after initiation
  at least 50% reduction in number of cigarettes smoked by week 16 of the intervention

SECONDARY OUTCOMES:
impact on inflammation -CRP | Mid of the intervention period 16 weeks after initiation
  Impact of smoking cessation/ reduction on inflammation measured with C-reactive protein in serum
impact on inflammation - leukocytes | Mid of the intervention period 16 weeks after initiation
  Impact of smoking cessation/ reduction on inflammation measured with total leukocyte count in blood
Number of cigarettes smoked | Mid of the intervention period 16 weeks after initiation
  If primary outcomes are not reached the daily number of cigarettes smoked is recorded
CO-levels in exhaled air | Mid of the intervention period 16 weeks after initiation
  If primary outcomes are not reached the CO levels in the exhaled air is recorded
Psychological distress | Mid of the intervention period 16 weeks after initiation
  Changes in psychological well-being will be assessed with the Norwegian validated translation ten item version of Hopkins Symptom Checklist (SCL-10)
Fatigue Symptom Scale | Mid of the intervention period 16 weeks after initiation
  Changes in fatigue will be assessed with the Fatigue Symptom Scale (FSS-3)
Physical functioning | Mid of the intervention period 16 weeks after initiation
  Physical functioning assessed with 4-minute step-test measuring number of steps climbed in period
Health-related quality of life | Mid of the intervention period 16 weeks after initiation
  Changes in health-related quality of life will be assessed with EuroQoL EQ-5D-5L
Health-related quality of life | Mid of the intervention period 16 weeks after initiation
  Changes in health-related quality of life will be assessed with self-reported question on happiness on a 0 to 10 scale

CONTACTS AND LOCATIONS:
Overall Officials: Lars Thore Fadnes, PhD, Principal Investigator — Haukeland University Hospital
Locations (2):
- Norway (2):
  - Department of Addiction Medicine, Haukeland University Hospital, Bergen
  - LAR Helse Stavanger HF, Stavanger

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Druckrey-Fiskaaen KT, Madebo T, Daltveit JT, Vold JH, Furulund E, Chalabianloo F, Gilje Lid T, Fadnes LT. Integrated Nicotine Replacement and Behavioral Support to Reduce Smoking in Opioid Agonist Therapy: A Randomized Clinical Trial. JAMA Psychiatry. 2025 Apr 1;82(4):406-414. doi: 10.1001/jamapsychiatry.2024.4801. PMID 39937506
- [Derived] Druckrey-Fiskaaen KT, Madebo T, Daltveit JT, Vold JH, Furulund E, Lid TG, Fadnes LT. Update of statistical analysis plan for: Integration of smoking cessation into standard treatment for patients receiving opioid agonist therapy who are smoking tobacco: protocol for a randomised controlled trial (ATLAS4LAR). Trials. 2024 Jan 6;25(1):29. doi: 10.1186/s13063-023-07894-w. PMID 38184633
- [Derived] Druckrey-Fiskaaen KT, Furulund E, Daltveit JT, Vold JH, Lid TG, Madebo T, Fadnes LT; ATLAS4LAR Study Group. Integration of smoking cessation into standard treatment for patients receiving opioid agonist therapy who are smoking tobacco: protocol for a randomised controlled trial (ATLAS4LAR). Trials. 2022 Aug 17;23(1):663. doi: 10.1186/s13063-022-06560-x. PMID 35978355
- See also: Project home page — https://helse-bergen.no/avdelinger/rusmedisin/rusmedisin-seksjon-forsking/bar/atlas4lar-kartlegging-og-behandling-av-lungesykdom-i-legemiddelassistert-behandling